CLINICAL TRIAL: NCT07137793
Title: Clinical Study to Evaluate The Cardioprotective Effect of Pentoxifylline Against Doxorubicin Induced Cardiotoxicity in Breast Cancer Patients
Acronym: PTX / BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sondos Mahmoud Elfeky, bachelor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TP/RE/5/25M-006
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Doxorubicin Induced Cardiotoxicity; Breast Cancer
Keywords: pentoxyfillne; breast cancer; cardioprotective; Doxorubicin Induced Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Pentoxifylline; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Positive control group receiving standard chemotherapy for breast cancer . (No Intervention)
- Pentoxifylline 400mg plus chemotherapy (Active Comparator)
  Interventions: Drug: Pentoxifylline 400mg plus chemotherapy

INTERVENTIONS:
Drug: Pentoxifylline 400mg plus chemotherapy — patient will receive standard chemotherapy for breast cancer plus pentoxifylline 400 mg orally 3 times per day with meals.
  Arms: Pentoxifylline 400mg plus chemotherapy

SUMMARY:
The goal of this clinical trial is to evaluate the cardioprotective effect of pentoxifylline against doxorubicin-induced cardiotoxicity in breast cancer patients. The main questions it aims to answer are:

1. What is the change in ejection fraction (primary outcome) in breast cancer patients receiving pentoxifylline compared to those who do not?
2. What are the changes in serum levels of N-terminal pro-B-type natriuretic peptide (NT-pro-BNP), and TNF-α (secondary outcomes) in breast cancer patients receiving pentoxifylline compared to those who do not? Researcher will compare breast cancer patients receiving standard chemotherapy alone (Group one: Positive control group; n=23) to breast cancer patients receiving standard chemotherapy plus pentoxifylline (Group two: pentoxifylline group; n=23) to see if pentoxifylline mitigates the cardiac side effects associated with doxorubicin treatment.

Participants will:

Be randomized to receive either a chemotherapeutic regimen alone or with pentoxifylline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Chemo-naïve patients with biopsy confirmed diagnosis of breast cancer and with stage I-III breast cancer according to the American Joint Committee on Cancer (TNM staging system of breast cancer).
* Patients intended to receive at least 4 cycles of doxorubicin or more.
* Patients with performance status <2 according to Eastern Cooperative Oncology Group (ECOG) score.
* Echocardiographic LVEF ≥55%.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 ×109/L, platelet count ≥ 90 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate liver function and adequate renal function.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years old and >65 years old.
* Women with history of breast cancer.
* Formerly treated with DOX.
* Patients with a known hypersensitivity to any of the used drugs.
* Treatment with blood thinners for 6 months prior to the screening.
* Treatment with NSAIDS like ketorolac,ibuprofen.
* Patients taking any other cardioprotective medications.
* Pregnancy and breast feeding.
* Alcohol abuse.
* Creatine Clearance < 50 mL/min.
* History of heart failure or LVEF <50%.
* Presence of any cardiac-related conditions such as angina pectoris, valvular disease, uncontrolled systemic hypertension, coronary heart disease, and cardiac surgery within the last 3 months.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females with breast cancer
Enrollment: 46 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
change in ejection fraction | 3 MONTHS

SECONDARY OUTCOMES:
changes in serum levels of the measured biological markers | 3 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Sahar kamal Hegazy professor, Study Chair — Tanta University; Eman Ibrahim Elberri Lecturer, Study Director — Tanta University
Locations (1):
- Damnhour Oncology Center, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matboli M, Habib EK, Hussein Mohamed R, Mahran NA, Seleem HS, Nosseir N, Hasanin AH. Pentoxifylline alleviated cardiac injury via modulating the cardiac expression of lncRNA-00654-miR-133a-SOX5 mRNA in the rat model of ischemia-reperfusion. Biomed Pharmacother. 2020 Apr;124:109842. doi: 10.1016/j.biopha.2020.109842. Epub 2020 Jan 20. PMID 31972363
- [Background] Dezube BJ, Sherman ML, Fridovich-Keil JL, Allen-Ryan J, Pardee AB. Down-regulation of tumor necrosis factor expression by pentoxifylline in cancer patients: a pilot study. Cancer Immunol Immunother. 1993;36(1):57-60. doi: 10.1007/BF01789132. PMID 7678547
- [Background] Fernandes JL, de Oliveira RTD, Mamoni RL, Coelho OR, Nicolau JC, Blotta MHSL, Serrano CV Jr. Pentoxifylline reduces pro-inflammatory and increases anti-inflammatory activity in patients with coronary artery disease--a randomized placebo-controlled study. Atherosclerosis. 2008 Jan;196(1):434-442. doi: 10.1016/j.atherosclerosis.2006.11.032. Epub 2006 Dec 28. PMID 17196208